CLINICAL TRIAL: NCT05116033
Title: Value of the Platelet Indices as a Predictive Factor in Adult Thrombocytopenic Patients
Brief Title: Value of Platelet Indices as Predictive Factor in Thrombocytopenia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahy nour Z Abed elhi,MD, Value of the platelet indices as a prognostic factor in adult thrombocytopenic patients, Assiut University
Other Study IDs: VOTIAAFITP
Record Dates: First submitted 2021-09-15; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Main Focus of the Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Platelets are essential blood component involved in primary hemostasis. A platelet count of less than 150 × 109/L is considered to be thrombocytopenia The causes of thrombocytopenia can be divided into two major groups, a decreased production of platelets or an under proliferative BM and an over-destruction of platelets. Under proliferative BM defects most common cause is aplastic anemia, On the contrary, peripheral destruction of platelets may be as a result of an immune-mediated process namely immune thrombocytopenia (ITP)

DETAILED DESCRIPTION:
ITP is a common auto-immune disease in which platelet count is reduced in peripheral blood leading to petechiae and hemorrhage. The platelet count is decreased because there are auto-antibodies in circulation against platelets that bind to platelets surface and destroy them in the spleen . Aplastic anemia is characterized by suppression of bone marrow function resulting in progressive pancytopenia. The hematology analyzers can now give us certain parameters that can give information about platelets. These parameters are referred to as platelet indices in literature. Platelet indices include mean platelet volume (MPV), platelet distribution width (PDW) and platelet large cell ratio (P-LCR) . They are sensitive, non-invasive, inexpensive biomarkers. MPV is the most commonly investigated platelet parameter, signifies the average size of platelets in the blood. PDW is a marker of platelet anisocytosis, which describes distribution of platelets produced by megakaryocytes and increases upon platelet activation. P-LCR is another marker of platelet activity, is a percentage of all platelets with a volume measuring over 12 fl circulating in the bloodstream .

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old regardless of gender.
* Platelet count below 100000/cu mm.
* Confirmed diagnosis aplastic anaemia.
* Confirmed diagnosis immune thrombocytopenia

Exclusion Criteria:

* Patient who received a platelet or blood transfusion within two weeks prior MPV analysis.
* Splenectomized patients
* Patients with chronic infection or inflammations.
* Diabetics and patients with coronary artery disease.
* Patients on anti- platelet or anti-inflammatory drugs.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants of the study will be confirmed as thrombocytopenic patients.
Sampling Method: Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2021-12-20 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the prognostic predictive value of the platelet indices in thrombocytopenic patients. | 6months
  • Exploring the validity of platelets indices as prognostic biomarkers in thrombocytopenic patients.

REFERENCES:
- [Result] Negash M, Tsegaye A, G/Medhin A. Diagnostic predictive value of platelet indices for discriminating hypo productive versus immune thrombocytopenia purpura in patients attending a tertiary care teaching hospital in Addis Ababa, Ethiopia. BMC Hematol. 2016 Jul 1;16:18. doi: 10.1186/s12878-016-0057-5. eCollection 2016. PMID 27375850
- [Result] Norrasethada L, Khumpoo W, Rattarittamrong E, Rattanathammethee T, Chai-Adisaksopha C, Tantiworawit A. The use of mean platelet volume for distinguishing the causes of thrombocytopenia in adult patients. Hematol Rep. 2019 Mar 29;11(1):7732. doi: 10.4081/hr.2019.7732. eCollection 2019 Feb 19. PMID 30996849
- [Result] Khan MI, Ullah I. Diagnostic importance of mean platelet volume, platelet distribution width and platelet large cell ratio as screening tool in immune thrombocytopenia. Porto Biomed J. 2020 Nov 24;5(6):e094. doi: 10.1097/j.pbj.0000000000000094. eCollection 2020 Nov-Dec. PMID 33283064
- [Result] Pogorzelska K, Kretowska A, Krawczuk-Rybak M, Sawicka-Zukowska M. Characteristics of platelet indices and their prognostic significance in selected medical condition - a systematic review. Adv Med Sci. 2020 Sep;65(2):310-315. doi: 10.1016/j.advms.2020.05.002. Epub 2020 Jun 4. PMID 32505856